CLINICAL TRIAL: NCT02837419
Title: A Multicenter Prospective Observational Cohort Study Determining the Cost-effectiveness of Extracorporal Life Support (ECLS) Treatment
Brief Title: Cost-effectiveness of Extracorporeal Life Support Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Willem Dieperink, research coordinator, University Medical Center Groningen
Other Study IDs: Dutch ECLS/2014/QoL
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Critically Ill
Keywords: extracorporeal life support; health related quality of life
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Health related Quality of life EQ-5D — Quality of Care

SUMMARY:
This study evaluates patients on ECLS treatment as considered appropriate with mortality and health related Quality of life and costs.

DETAILED DESCRIPTION:
A direct comparison between usual care and ECLS treatment is difficult. Alternatively we compare predicted mortality for every patient based on validated scoring systems at the initiation of ECLS treatment with the actual outcome, so every patient is his own control.

Primary outcome is HRQoL assessed with the EQ-5D questionnaire at 1 year. Healthcare costs and costs from a societal perspective are prospectively measured.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care
* Treated with extracorporeal life support

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients on the ICU treated with extracorporeal life support
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
health related quality of life | 12 months
  health related quality of life with EQ-5D questionnaire at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: walter m van den Bergh, MD, PhD, Principal Investigator — department of critical care, UMCG
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Jolink FEJ, Onrust M, Dos Reis Miranda D, Mandigers L, Delnoij T, Maas JJ, Raasveld SJ, Vlaar APJ, Donker DW, Scholten E, de Metz J, van den Brule J, Kuijpers M, Vermeulen KM, van der Voort PHJ, van den Bergh WM, Oude Lansink-Hartgring A; Dutch Extracorporeal Life Support (ECLS) Study Group. Five Years After Extracorporeal Membrane Oxygenation: A Prospective Cohort Study of Health-Related Quality of Life and Patient Outcomes. Crit Care Med. 2025 Dec 1;53(12):e2487-e2496. doi: 10.1097/CCM.0000000000006900. Epub 2025 Oct 15. PMID 41091003
- [Derived] Oude Lansink-Hartgring A, Dos Reis Miranda D, Donker DW, Maas JJ, Delnoij T, Kuijpers M, van den Brule J, Scholten E, Endeman H, Vlaar APJ, van den Bergh WM; Dutch ECLS study group. Cost-effectiveness in extracorporeal life support in critically ill adults in the Netherlands. BMC Health Serv Res. 2018 Mar 9;18(1):172. doi: 10.1186/s12913-018-2964-6. PMID 29523153